CLINICAL TRIAL: NCT02992860
Title: Single Agent JNJ-56022473 in MDS and AML Patients Failing Hypomethylating Agent Based Therapy
Acronym: SAMBA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollement was stopped due to a recommendation by the IDMC/FDA for a parallel clinical trial with TALA, where potentielly no efficancy could be determined.
Sponsor: GWT-TUD GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAMBA-trial; 11274 (Other: GWT-TUD GmbH)
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Myelodysplastic Syndrome (MDS); Acute Myeloid Leukemia (AML)
Keywords: Myelodysplastic Syndrome (MDS); Acute Myeloid Leukemia (AML); hypomethylating agent (HMA) treatment; leukemic stem cell; CD123; immunotherapy
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Blood Cell Count; Cytogenetic Analysis; Pregnancy Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): JNJ-56022473 will be given intravenously to all subjects at a dose of 9 mg/kg once every 14 days for an initial treatment period of 3 months (6 infusions). Responders will then receive up to 20 additional infusions whereas for non-responders the initial treatment will be followed by a up to 9 months observation period without further JNJ-56022473 treatment. Thus, the individual study duration for a subject will be approx. 1 year. A follow up visit will be performed after 3 months after last study drug administration for all patients to track pregnancy status according to IB.
  Interventions: Drug: JNJ-56022473; Procedure: Bone marrow analyses and CBC with differential; Other: Flow cytometry analyses; Other: Central biobanking; Procedure: Histopathology analysis; Genetic: Cytogenetic analysis; Procedure: Serum chemistry; Procedure: Automated CBC; Procedure: Pregnancy Test

INTERVENTIONS:
Drug: JNJ-56022473 — JNJ-56022473 will be supplied as a lyophilized product containing 100mg of active pharmaceutical ingredient (50 mg/mL after reconstitution with 2.0 mL sterile water for injection). The JNJ-56022473 dose administered will be dependent upon the subject's weight at baseline. The JNJ-56022473 dose should be adjusted in case the subject's weight changes by > 10%. JNJ- 56022473 will be administered in 250 mL IV infusion over approximately 180 minutes using an infusion pump.
  Other Names: CSL362
Procedure: Bone marrow analyses and CBC with differential — Bone marrow analyses and CBC with differential will be performed by a central laboratory. If the marrow cannot be aspirated, a biopsy should be performed.
Other: Flow cytometry analyses — Characterization of LSCs and blasts (including CD123 and CD38 expression) will be performed as study-related analyses in the context of this protocol by central flow cytometry using bone marrow samples.
Other: Central biobanking — Central biobanking of study samples (bone marrow, peripheral blood as well as a buccal swab) will be carried out in Dresden.
Procedure: Histopathology analysis — A bone marrow biopsy is taken whenever it seems necessary to the investigator.
Genetic: Cytogenetic analysis — The cytogenetic analysis with banding analysis (optional FISH) have to be performed at local labs. Therefore 2 - 5 ml of bone marrow will be collected and analysed.
Procedure: Serum chemistry — For serum chemistry 15 ml (2 x 7,5 ml) of peripheral blood have to be collected.
Procedure: Automated CBC — For CBC a minimum of 3 ml of peripheral blood have to be collected.
Procedure: Pregnancy Test — Serum or urine pregnancy testing β-HCG with a sensitivity of at least 25 mIU/mL is to be done not more than 3 days prior to initiation of JNJ-56022473 in female patients with childbearing potential. Furthermore, serum or urine pregnancy testing has to be done after end of treatment (EoT) visit.

SUMMARY:
The outcome of HMA-refractory patients with MDS or AML is dismal with a median survival of 5 months after failure, representing a significant unmet medical need due to the very limited treatment options. In this context, a specific targeting of the leukemic stem cell (LSC) seems a promising option to selectively combat the leukemic progenitor cells. In fact, CD123 is overexpressed in AML and MDS progenitors making it an attractive target for immunotherapy-based approaches. JNJ-56022473 is a promising compound that has been engineered with regard to this strategy and the current phase II trial has the aim to evaluate the overall hematological response rate at 3 months in HMA refractory/relapsed AML and MDS patients.

DETAILED DESCRIPTION:
Myelodysplastic syndromes (MDS) comprise a heterogeneous group of hematologic malignancies of the pluripotent hematopoietic stem cells characterized by clonal hematopoiesis and progressive bone marrow failure. Clinically, patients suffer from fatigue and are at high risk of infections or bleeding. Also, MDS patients are endangered by progression to secondary acute myeloid leukemia (AML), a disorder of early hematopoietic progenitor cells characterised by the clonal expansion of myeloid blasts in the peripheral blood, bone marrow, and/or other tissues.

Up to now, allogeneic transplantation is considered the only curative option for both MDS and AML patients. However, as MDS and AML mainly manifest in the 7th and 8th decade of life, only a limited number of patients tolerating bone marrow transplantation and are therefore eligible for this procedure. In fact, comorbid conditions are common among the elderly such as heart disease, renal insufficiency and vascular disease thus influencing the ability to withstand exhausting transplantation procedures.

Hence in recent years, novel therapeutic strategies have been developed and hypomethylating agents (HMAs) azacitidine and decitabine have emerged as new therapeutic options. In 2009, azacitidine was the first HMA in use having received approval for treatment of MDS and AML patients with 20-30% blasts. In 2012, also the sister compound decitabine got approval for treatment of AML patients ≥ 65 years of age and in 2015, azacitidine's approval was extended to AML patients ≥ 65 years of age that are considered unfit for allogeneic transplantation with > 30% blasts.

However, despite the efficacy and reported activity, only 50% of patients respond to the treatment with HMAs and the majority of them do relapse. Also the outcome of HMA- refractory patients is dismal with a median survival of 5 months after failure and hence MDS and AML patients with HMA failure represent a significant unmet medical need due to the poor prognosis and very limited treatment options.

In this context, a specific targeting of the leukemic stem cell (LSC) seems a promising option to selectively combat the leukemic cells. In fact, CD123 (also known as interleukin-3-Rα) is expressed in different hematological malignancies, among others in MDS and AML. Interestingly, CD123 is expressed by the majority of AML blasts and it is also overexpressed by CD34+ CD38- LSCs compared with normal hematopoietic stem cells and other normal tissues. These features make CD123 an attractive target for anti-leukemia therapy. Recent data suggests that treatment with HMA can induce expression of CD123 on AML tumors opening up the potential that HMA failure patients may have even higher expression levels of CD123.

Indeed, JNJ-56022473 is a promising compound that has been engineered with regard to this strategy. JNJ-56022473 is a humanized monoclonal antibody that targets the alpha chain of the interleukin-3-receptor and is optimized at the Fcγ region for enhanced activation of antibody- dependent cell-mediated cytotoxicity (ADCC) via natural killer cells.

Recently, JNJ-56022473 has been evaluated in a phase I study with AML patients at high risk for early relapse. There was a clear dose dependency on depletion of peripheral CD123 cell populations such as pDC and basophile with complete and sustained depletion seen in pts at doses ≥3 mg/kg Given the encouraging results of this phase I trial we now propose a phase II trial to evaluate JNJ-56022473 in AML patients as well as in MDS patients that have failed or are refractory to HMA- treatment.

The clinical trial will be accompanied by a translational research program which aims at elucidating specific immune responses mediated by JNJ-56022473, in particular by descriptive and functional analyses. In this context bone marrow and peripheral blood will be collected during the study as well as before and after therapy.

Constitutive overexpression of the α-subunit of the interleukin-3 receptor i.e. IL-3Rα, is a hallmark of the early AML progenitor cell population (i.e. leukemic stem cells) as well as leukemic blasts and IL-3Rα is also overexpressed in myelodysplastic syndromes. In fact, CD123 is unique to the IL-3 receptor and is responsible for the high specificity and low affinity binding of IL-3. Upon ligand binding, the α-subunit CD123 associates with the βc-subunit (CD131) to form a high-affinity receptor complex initiating an intracellular signaling cascade through phosphorylation and activation of at least 3 distinct signal transduction pathways: the JAK/STAT-kinase, MAP-kinase-, and PI3-kinase-pathways. Under physiological conditions, activation of the IL-3 receptor induces proliferative, anti-apoptotic, and differentiating signals.

JNJ-56022473 (CSL362) is a second generation antibody developed from the murine 7G3 anti- CD123 monoclonal antibody (mAb) in a stepwise process of humanization, affinity maturation, and Fc engineering. To enhance the cytotoxicity of the first-generation antibody CSL360, the proprietary Xencor (Xmab®) technology was applied and two amino acid mutations (S239D and I332E) were introduced into the Fc region. These amino acid substitutions led to improved binding to CD16 (FcγRIIIa) on natural killer (NK) cells and significantly enhanced the ability to induce ADCC.

The JNJ-56022473 drug product that will be used in this study is produced in a different cell line with a different process compared with CSL362, the drug product used in the phase I study CSLCT-AML-11-73 described below. Comparability testing of JNJ-56022473 and CSL362 has shown the antibodies to behave similarly in biophysical, biochemical, and preclinical assessments. The primary structure, charge heterogeneity, size heterogeneity, purity, higher order structure, and process impurities were found to be highly similar between CSL362 and JNJ56022473. Pharmacodynamic (PD) studies in cynomolgus monkeys showed similar levels of biological activity between CSL362 and JNJ-56022473 (ie, basophil and pDC depletion; NK cell number and activity). Additionally, the pharmacokinetic (PK) profiles of JNJ-56022473 following 30 and 100 mg/kg IV dosing of cynomolgus monkeys are highly similar to those of CSL362. Following the first weekly intravenous dose, mean Cmax and AUC0-167h of JNJ-56022473 are 91% and 94% of those observed for CSL362, respectively.

This is an open-label, single-arm, multicenter, phase II study of JNJ-56022473 in subjects suffering from MDS or AML. The trial will involve participating sites from Germany and France. Up to a maximum of 43 subjects will be enrolled in the study.

JNJ-56022473 will be given intravenously to all subjects at a dose of 9 mg/kg once every 14 days for an initial treatment period of 3 months (6 infusions). Responders will then receive up to 20 additional infusions whereas for non-responders the initial treatment will be followed by a up to 9 months observation period without further JNJ-56022473 treatment. Thus, the individual study duration for a subject will be approx. 1 year. A follow up visit will be performed after 3 months after last study drug administration for all patients to track pregnancy status according to IB.

For patients who still benefit from the treatment and are graded as responders after the time period defined above, treatment will continue as long as medically indicated. End of study as a whole will be 16 months after LPFV (maximum of 26 treatment cycles plus follow up of three months). Data obtained after the end of the study (EoS) for patients who still responding will be reported under separate cover.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Diagnosis of AML or MDS
* At least ≥ 5% BM blasts at the time of screening (done by central morphology)
* At least one cytopenia (ANC < 1800/μL or platelet count < 100,000/μL or hemoglobin < 10 g/dL)
* Failure to achieve complete or partial response or hematological improvement after at least six (azacitidine) or four (decitabine) 4-week treatment cycles administered during the past two years OR
* Relapse after initial complete or partial response or hematological improvement observed after at least six (azacitidine) or four (decitabine) 4-week treatment cycles administered during the past two years OR
* Intolerance to treatment with HMA (hypomethylating agents) defined by drug-related ≥ Grade 3 liver or renal toxicity leading to treatment discontinuation during the past two years
* Failed to respond to, relapsed following, not eligible, or opted not to participate in bone marrow transplantation
* Off all other treatments for AML/MDS for at least four weeks; Filgrastim (G-CSF) and erythropoietin are allowed before and during the study as clinically indicated
* No medical need for or patient opted not to receive induction chemotherapy
* ECOG performance status of 0-2
* Willing to adhere to the prohibitions and restrictions specified in the protocol
* Signed informed consent

Exclusion Criteria:

* Previous treatment with a CD123 agent or T- or NK cell redirecting therapy
* Patients having received intensive chemotherapy to treat HMA failure
* Diagnosis of acute promyelocytic leukemia (APL)
* WBC > 15 GPT/L
* Any active malignancy within the past year, except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or breast
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
* Active infection not adequately responding to appropriate therapy
* Total bilirubin > 1.5 mg/dL not related to hemolysis or Gilbert's disease
* ALT/AST > 2.5 x upper limit of normal
* Serum creatinine > 2.0 mg/dL
* Patients who are unwilling to follow highly effective contraception requirements (including condom use for males with sexual partners, and for females: prescription oral contraceptives, contraceptive injections, intrauterine device, , contraceptive patch, surgical sterilization or true sexual abstinence) before entry, at least at screening, throughout the study and within 3 months after last study drug administration
* Female patients with reproductive potential who do not have a negative urine β-HCG pregnancy test at screening and prior to the first study drug administration at visit 1 (day 0) of JNJ-56022473 treatment period.
* Female patients who are lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Overall hematological response rate | 3 months
  Overall hematological response rate at 3 months (either CR, PR, marrow-CR, HI, SD)

SECONDARY OUTCOMES:
Toxicity | 3 or 12 months
  Toxicity as measured by NCI CTCAE 4.03
Overall survival | 1 year
Progression-free-survival | 1 year
Overall hematological response rate at 12 months | 1 year
Quality of life EORTC-QLQ30 | 9 or 15 months
  measured by EORTC-QLQ30
Time to treatment failure | 3 or 12 months
Duration of response (best overall response) | 3 or 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Platzbecker, Prof., Principal Investigator — Universitätsklinikum Dresden; Lionel Adés, Dr., Principal Investigator — Hospital Saint Louis Paris
Locations (10):
- France (4):
  - CHU Nantes, Nantes
  - Hospital Archet 1, Nice
  - Hospital Saint Louis, Paris
  - CHU Toulouse, Toulouse
- Germany (6):
  - Klinikum Chemnitz gGmbH, Klinik für innere Medizin III, Chemnitz
  - Universitätsklinikum Dresden, Dresden
  - Heinrich Heine Universität, Düsseldorf
  - Marien Hospital GmbH, Düsseldorf
  - Technische Universität München, Klinikum rechts der Isar, Munich
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No